CLINICAL TRIAL: NCT04088877
Title: Restoring Body Image After Breast Cancer Through Exercise and Art Sculpture "RISE UP" After Breast Cancer: A Pilot Multi-Methods Study
Brief Title: Rise Up After Breast Cancer
Acronym: RISE-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC 19-0363
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Body Image
Keywords: Exercise; Art sculpture; Breast neoplasms; Body Image
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Masking Description: Independent assessors will assess outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise and Art Sculpting Class (Experimental): Participants will take part in a twelve week exercise program twice per week as well as an eight week art sculpting class once a week.
  Interventions: Behavioral: Exercise; Behavioral: Art Sculpting Class

INTERVENTIONS:
Behavioral: Exercise — The participants will attend the exercise facility at Wellspring two times a week. Sessions are completed under the supervision of an exercise physiologist and the duration of each session ranges from 1.0 - 1.5 hours. Each session includes a warm up on an aerobic exercise machine, a full body progressive RET program followed by balance and stretching exercises.
Behavioral: Art Sculpting Class — The sculpting program will take place once a week for 2 hours over an 8-week period. Sessions will be themed around body image and facilitated by an artist and registered psychologist who will lead the group in art techniques and self-reflection, respectively. Each group session will focus on a theme related to body image, and the participants will have the opportunity to reflect through their art and social interactions with one another.

SUMMARY:
The objectives of this pilot study are to determine the feasibility of a community-based moderate intensity resistance exercise training (RET) program in combination with an art sculpting class on body image in breast cancer survivors (BCS). The protocol will be measuring recruitment; attendance; cost tracking; body image distress; body image appreciation; and muscular strength. Participant feedback on the intervention will be collected through a final focus group. Additionally, cognitive interviews will occur prior to the intervention, where participants will be asked to "think-out-loud" as they answer the Body Image Scale for Cancer questionnaire. The purpose of this interview technique is to gain a deeper understanding of the participants' thought process behind choosing each answer. The proposed pilot study will be a single prospective before and after study that will help inform a future large-scale project. A minimum sample of 12 subjects will be recruited.

The Health Research Ethics Board of Alberta Cancer Committee will approve this study. Participants will participate in RET biweekly for 12 weeks and the sculpting class weekly for 8 weeks. After the first week of RET, the art class will begin. Both the RET and sculpting class will be between 1-2 hours in length.

Analyses: Quality of life, fitness testing and body image scales will be administered before and after the intervention. Cognitive interviews will occur once before the intervention has started and a final focus group will occur at the end of the intervention to get participant feedback on the effectiveness of the program

DETAILED DESCRIPTION:
Breast cancer is the third most frequently diagnosed cancer in Canada. Treatment of breast cancer typically involves an initial surgery, followed by radiation, chemotherapy and hormonal treatments. These treatments are invasive and may result in a visible change in a survivor's physical appearance, which can lead to body image concerns, depression, and psychological distress. Currently, many of the studies that address body image in breast cancer use a biomedical model, often ignoring the need for incorporating behavioural and psychosocial aspects of the construct.

Resistance exercise training (RET) holds promise as an intervention to help improve body image among women in the general population. Art classes have been found to have a positive impact on cancer survivors' psychological and spiritual well-being, quality of life, and coping. To date, however, the evidence is limited regarding interdisciplinary approaches to addressing body image in breast cancer. This study will examine the feasibility and preliminary efficacy of combining a resistance exercise training program with a group art sculpting class to address body image in breast cancer.

The main objectives of this project are: 1) To determine the feasibility and preliminary efficacy of a RET program and art sculpting class on body image in breast cancer survivors.

2) Determine if the Body Image Scale for Cancer (BIS) survey reflects the experiences breast cancer survivors have with their body image.

3) Evaluate the patient experience through a final focus group This study will be a prospective before and after pilot study with baseline measures that include: collection of participant demographics, quality of life, baseline fitness tests, body image scales, and cognitive interviews. After the intervention, the following measures will be collected: quality of life, fitness tests, body image scales, recruitment/adherence data, and intervention feedback through a final focus group.

A minimum sample of 12 subjects who previously attended the Alberta Cancer Exercise program (ACE) in Edmonton will be recruited for this project. Subjects will be screened for eligibility and if they meet all eligibility criteria, an information letter of the study will be provided and they will be asked to contact the investigators if interested in taking part in the study. All participant will be required to provide signed informed consent as per the Health Research Ethics Board (HREB) of Alberta: Cancer Committee.

Participants will participate in a 12-week resistance exercise program, twice a week and an Art Sculpting class for 8-weeks. From week 2 to 10 of the intervention, the group art sculpting class take place once a week. Both the exercise and art classes will take place at Wellspring Edmonton, a non-profit community center that provides supportive Wellness programming for cancer survivors.

RET: The participants will attend the exercise facility at Wellspring two times a week. Sessions are completed under the supervision of an exercise physiologist and the duration of each session ranges from 1.0 - 1.5 hours. Each session includes a warm up on an aerobic exercise machine, a full body progressive RET program followed by balance and stretching exercises.

Art Sculpting Class: The sculpting program will take place once a week for 2 hours over an 8-week period. Sessions will be facilitated by an artist and registered psychologist who will lead the group in art techniques and self-reflection, respectively. Each group session will focus on a positive health theme related to body image, and the participants will have the opportunity to reflect through their art and social interactions with one another.

Statistical Analysis: Demographic and medical information will be presented using median and range and percentage for interval and nominal data respectively. The primary analysis will compare outcomes before and after the intervention with regard to body image perception from the survey tools and the fitness testing results. This will meet the preliminary efficacy objectives of the study; to determine whether the intervention demonstrates a trend towards improved body image. Analyses of outcomes will be performed at the end of the intervention using non-parametric tests (Wilcoxon signed rank). Point estimates and measures of variability to inform future research will be calculated from parametric statistics using a paired t-test.

Qualitative Analysis: Qualitative data will be collected at two separate time points - once, through the cognitive interviewing of the BIS scale and the second through the focus group at the end of the intervention. An abductive analytical approach using a semantic analysis from Braun and Clarke (2006) will be used to understand the various participant perspectives and contextualize the participants' experiences. The methodology used for the cognitive interviewing will be interpretive description.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age and older;
2. Diagnoses of breast cancer stage I-III;
3. Identify issues with body image on the Alberta Cancer Exercise intake form
4. Cleared for unrestricted physical activity by the Certified Exercise Physiologist on the PAR-Q+
5. Participants must have completed their cancer treatments
6. Participants must have completed the Alberta Cancer Exercise 12-week program

Exclusion Criteria:

1. Presence of active cancer or metastatic disease;
2. Serious or uncontrolled co-morbid disease or injury that would be deemed unsafe to exercise (e.g. Uncontrolled diabetes, heart failure);
3. Has undergone breast reconstruction surgery;
4. Inability to provide consent;
5. Inability to commit to, and/or comply with the intervention due to personal reasons (e.g. vacation planned during the intervention period)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Completion rate | 12-weeks
  Number of participants starting the study divided by the number enrolled

SECONDARY OUTCOMES:
Recruitment rate | 12-weeks
  Number of participants enrolling in the study divided by the number eligible
Adherence rate | 12-weeks
  Participant adherence at schedule exercise and art class sessions
Body Image Scale (BIS) | 12-weeks
  Change in body image: 10-item scale: body image symptoms are scored on a 4-point scale (0 "not at all" to 3 "very much"). The total score ranges from 0 to 30 and can be calculated by summing up the 10 items. A higher score means a higher level of body image disturbance.
Body Appreciation Scale- 2 (BAS-2) | 12-weeks
  Body Appreciation Scale Version 2: This is a 10-item questionnaire: body appreciation is scored on a 5-point scale with 1 (never) to 5 (always) related to each question. Full scale is scored out of 50, with higher scores indicating higher body appreciation.
Patient Experience | 12-weeks
  Focus group session: qualitative
One repetition maximum strength upper body | 12-weeks
  Vertical bench: one repetition maximum test
One repetition maximum strength lower body | 12-weeks
  Leg press: one repetition maximum test
Functional Assessment of Cancer Therapy: Fatigue Sub-scale | 12-weeks
  Symptoms of Fatigue: scored out of 52 points with higher scores indicating less fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF